CLINICAL TRIAL: NCT01446939
Title: Role of Diffusion Tensor Imaging and Transcranial Sonography in the Parkinson's Disease and Essential Tremor
Brief Title: Imaging in the Diagnosis of Parkinson's Disease and Essential Tremor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ellison Fernando Cardoso, MD, PhD, Hospital Israelita Albert Einstein
Other Study IDs: IIEP1436-11; CAPPESQ8197 (Other: Faculdade de Medicina da Universidade de São Paulo)
Record Dates: First submitted 2011-09-13; First posted 2011-10-05 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson's Disease; Essential Tremor
Keywords: MRI; Parkinson's disease; Essential tremor; Ultrasonography; Diagnosis
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Parkinson's disease: Patients with primary Parkinson's disease
- Essential tremor: Patients with essential tremor
- Healthy volunteers: Healthy volunteers

SUMMARY:
Parkinson´s disease (PD) diagnosis is based upon clinical examination. Although imaging has helped doctors to identify many diseases, it still does not add too much information for the diagnosis of Parkinson´s disease. The investigators are going to perform a large sample study including PD patients, essential tremor and healthy volunteers in order to evaluate if MRI can help in the diagnosis. Our hypothesis is that fractional anisotropy (FA) in the caudal portion of substantia nigra is decreased in PD patients.

DETAILED DESCRIPTION:
The diagnosis of Parkinson's disease (PD) is based on a set of clinical assessments that do not provide great accuracy. Although magnetic resonance imaging (MRI) and transcranial sonography (TCS) have provided important advances in the diagnosis of a number of neurological diseases, few biomarkers of PD have been described in order to support its clinical diagnosis.

Recently, one single study showed that high field MRI using diffusion tensor imaging (DTI) was able discriminate PD from healthy volunteers. This study had a small sample size (14 patients and 14 controls) and did not include the main differential diagnosis of PD.

The main objective of this study is to confirm previous findings, with a larger sample size, describe possible changes of DTI parameters in patients with essential tremor (one of the main differential diagnosis of PD), and compare DTI MRI with TCS. Our primary outcome will be the fractional anisotropy (FA) in the caudal portion of substantia nigra. As a consequence, new algorithm to discriminate PD, essential tremor and healthy volunteers will be proposed. This has a pivotal importance in order to provide support to clinical diagnosis of PD and increase its accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson´s disease patients according to UK Parkinson´s Disease Brain Bank Criteria
* Essential Tremor Patients according to Movement Disorder´s diagnosis consensus criteria.
* Healthy Volunteers: paired with PD patients by age and gender.

Exclusion Criteria:

* Contraindication to MRI
* Claustrophobia.
* Serious structural brain anomalies.
* Condition or situation in which, in the opinion of the investigator put the patient at significant risk, which can confound the results, or substantially interfere with the individual's participation in the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 Parkinson´s Disease Patients 50 Essential Tremor Patients 50 Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-02 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Fractional anisotropy (FA) in the caudal portion of substantia nigra | baseline (MRI study date)
  Fractional anisotropy (FA) in the caudal portion of substantia nigra.

SECONDARY OUTCOMES:
Comparison between MRI and ultrasonography | baseline (Date of ultrasonography)
  Comparison between MRI and ultrasonography in the accuracy of diagnosis through ROC curves

CONTACTS AND LOCATIONS:
Overall Officials: Edson Amaro Junior, MD,PhD, Study Chair — Hospital Israelita Albert Einstein; Claudia C Leite, MD, PhD, Study Chair — Faculdade de Medicina da Universidade de São Paulo
Locations (2):
- Brazil (2):
  - Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo

REFERENCES:
- [Background] Vaillancourt DE, Spraker MB, Prodoehl J, Abraham I, Corcos DM, Zhou XJ, Comella CL, Little DM. High-resolution diffusion tensor imaging in the substantia nigra of de novo Parkinson disease. Neurology. 2009 Apr 21;72(16):1378-84. doi: 10.1212/01.wnl.0000340982.01727.6e. Epub 2009 Jan 7. PMID 19129507